CLINICAL TRIAL: NCT00068367
Title: U.S./Canada Sarcoma Intergroup Study of OSI-774 in Malignant Peripheral Nerve Sheath Tumors, Phase II
Brief Title: S0330 Erlotinib in Treating Patients With Unresectable or Metastatic Malignant Peripheral Nerve Sheath Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000322023; S0330 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Sarcoma
Keywords: adult neurofibrosarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Neurofibrosarcoma | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (OSI-774) (Experimental): Drug: erlotinib hydrochloride
  Other Names:
  OSI-774 150 mg per day, daily until disease progression
  Interventions: Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — 150 mg per day, daily until disease progression
  Other Names: OSI-774

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with unresectable or metastatic malignant peripheral nerve sheath tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response (confirmed, complete, and partial) in patients with unresectable or metastatic malignant peripheral nerve sheath tumor when treated with erlotinib.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Correlate, preliminarily, indicators of epidermal growth factor receptor (EGFR) function (e.g., expression, phosphorylation, or markers of signal transduction downstream of EGFR) with response and progression-free and overall survival in patients treated with this drug.
* Determine the feasibility of accruing these patients in the cooperative group setting.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients who achieve at least a confirmed partial response and become resectable undergo surgical resection (with or without radiotherapy) and then receive 2 additional courses of erlotinib. Patients with responding disease who do not become resectable continue erlotinib as above. Patients achieving a complete response (CR) receive 2 additional courses of erlotinib beyond the CR.

Patients are followed every 6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant peripheral nerve sheath tumor

  * Malignant schwannoma or neurofibrosarcoma
  * Clinical evidence of unresectable or metastatic disease
* Measurable disease
* No known current CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 1.5 times ULN (5 times ULN for patients with documented liver metastases)

Renal

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance greater than 60 mL/min

Ophthalmic

* No known history of any of the following corneal diseases:

  * Dry eye syndrome
  * Sjögren's syndrome
  * Keratoconjunctivitis sicca
  * Exposure keratopathy
  * Fuch's dystrophy
* No other active disorders of the cornea

Gastrointestinal

* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No active peptic ulcer disease
* No intractable nausea or vomiting
* Able to swallow medications OR receive enteral medications via gastrostomy feeding tube

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy for this malignancy

Chemotherapy

* More than 28 days since prior chemotherapy for this malignancy

Endocrine therapy

* Not specified

Radiotherapy

* More than 60 days since prior radiotherapy to the target lesion with subsequent documented progression
* More than 60 days since prior radiofrequency ablation to the target lesion with subsequent documented progression
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior major surgery and recovered
* No prior surgical procedure affecting absorption

Other

* More than 28 days since prior investigational drugs for this malignancy
* More than 60 days since prior embolization to the target lesion with subsequent documented progression
* No prior epidermal growth factor receptor-targeting therapy
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-12; Primary Completion 2007-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Albritton, MD, Study Chair — Dana-Farber Cancer Institute; R. Lor Randall, MD, FACS, Study Chair — University of Utah; Scott M. Schuetze, MD, PhD, Study Chair — University of Michigan Rogel Cancer Center
Locations (101):
- United States (101):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Davis Cancer Center, Davis, California
  - Contra Costa Regional Medical Center, Martinez, California
  - St. Anthony Central Hospital, Denver, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - St. Anthony North Hospital, Westminster, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Piedmont Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Danville Regional Medical Center, Danville, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Regional Cancer Center at Providence Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Albritton KH, Rankin C, Coffin CM, et al.: Phase II study of erlotinib in metastatic or unresectable malignant peripheral nerve sheath tumors (MPNST). [Abstract] J Clin Oncol 24 (Suppl 18): A-9518, 524s, 2006.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four patients enrolled to study were found to be ineligible. One patient did not have measurable disease, one patient had radiotherapy 19 days prior to registration and two patients were found ineligible upon pathology review.
Groups:
- Arm I (OSI-774): OSI-774 150 mg daily for 25 weeks
Period: Overall Study
Arm/Group | Arm I (OSI-774)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I (OSI-774)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 45.3 [19.8 to 76.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Prior multi-agent chemotherapy [Count of Participants; unit: Participants]
  Yes | 14
  No | 6

OUTCOME MEASURES:

1. Primary Outcome: Patients With Response (Confirmed Complete, and Partial) With Unresectable or Metastatic Malignant Peripheral Nerve Sheath Tumor When Treated With Erlotinib.
Description: Complete response - Complete disappearance of all measurable and non-measurable disease. No new lesions, no disease related symptoms, normalization of markers and other abnormal lab values.
  Partial response - Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease, no new lesions.
Time Frame: 25 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (OSI-774)
Number analyzed (Participants) | 20
Participants | 0

2. Secondary Outcome: Toxicity
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 25 weeks
Population: All participants receiving at least some protocol treatment
Measure: Number; unit: Participants
Arm/Group | Arm I (OSI-774)
Number analyzed (Participants) | 20
Participants
  Anorexia | 1
  Diarrhea | 1
  Dyspnea (shortness of breath) | 1
  Fatigue (asthenia, lethargy, malaise) | 3
  Hemoglobin | 1
  Nausea | 1
  Pain - Abdomen NOS | 1
  Pruritus/itching | 1
  Rash/desquamation | 1
  Somnolence/depressed level of consciousness | 1
  Vision-blurred vision | 1

3. Other Pre Specified Outcome: Correlate, Preliminarily, Indicators of Epidermal Growth Factor Receptor (EGFR) Function With Response and Progression-free and Overall Survival in Patients Treated With This Drug.
Description: NOT COMPLETED DUE TO EARLY CLOSURE OF STUDY
Arm/Group | Arm I (OSI-774)
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Feasibility of Accruing These Patients in the Cooperative Group Setting
Description: NOT COMPLETED DUE TO EARLY CLOSURE OF STUDY
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 25 weeks
Arm/Group | Arm I (OSI-774)
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (OSI-774) (N=20)
Diarrhea (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (OSI-774) (N=20)
Hemoglobin (Blood and lymphatic system disorders) | 2
Dry eye syndrome (Eye disorders) | 1
Ocular/Visual-Other (Eye disorders) | 2
Vision-blurred vision (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 1
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Edema: head and neck (General disorders) | 1
Edema: limb (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 2
Pain - Chest/thorax NOS (General disorders) | 1
Pain-Other (General disorders) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 1
Lymphopenia (Investigations) | 2
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 3
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dizziness (Nervous system disorders) | 1
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Ocular/Visual-Other (Nervous system disorders) | 2
Pain - Head/headache (Nervous system disorders) | 4
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Mood alteration - depression (Psychiatric disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hemorrhage/Bleeding-Other (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less